CLINICAL TRIAL: NCT03409029
Title: A Pilot Study Using Magnetic Resonance Imaging (MRI) to Assess Bladder Motion During Radiotherapy Treatment.
Brief Title: A Study Using MRI To Assess Bladder Motion During Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sally Falk, Research Project Manager, The Christie NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17_RADIO_130
Record Dates: First submitted 2018-01-10; First posted 2018-01-24 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Bladder Cancer
Keywords: bladder; radiotherapy; magnetic resonance imaging
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Single site, non-randomised basic science study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI Scan (Experimental): As part of the study patients will undergo 4 MRI scans during radiotherapy treatment. These will take place during the 1st, 2nd, 3rd and 4th week of treatment
  Interventions: Diagnostic Test: MRI Scan

INTERVENTIONS:
Diagnostic Test: MRI Scan — Additional imaging using MRI scan

SUMMARY:
The standard non-surgical treatment for muscle invasive bladder cancer is concurrent chemo-radiotherapy. This treatment is associated with long term side effects in around a third of patients with up to 12% suffering from grade 3-4 toxicity.

Effective radiotherapy depends on delivering a curative dose to the target whilst minimising dose to surrounding tissues to reduce toxicities. As an organ that constantly varies in shape and position, achieving this in bladder irradiation is challenging. Cone beam Computed Tomography (CBCT) has allowed visualisation of soft tissue on treatment and hence image-guided treatment and improved accuracy, but the image quality of CBCT is suboptimal for distinguishing soft tissue boundaries. On the other hand, MRI scans produce superior soft tissue definition and visualisation of tumour bed. This would in turn allow for various ways of optimising treatment and potentially improving outcome.

There have been a number of studies evaluating pelvic organ motion in bladder cancer as well as assessing different adaptive radiotherapy strategies. These have included individualized margins, plan of the day and adaptive techniques. Most of these studies have been carried out using CBCT imaging which is often poor quality with limited soft tissue contrast. MRI offers better visualization of the tumour bed and organs at risk (OARs). As a result, the utilisation of MRI in radiotherapy could allow for increased radiation dose to the tumour bed while maintaining minimal dose to surrounding soft tissue.

This study will explore the role of MRI imaging in adaptive radiotherapy for bladder cancer with development of a number of theoretical treatment strategies.

DETAILED DESCRIPTION:
Patients will undergo standard treatment during the study with four weeks of external beam radiotherapy (20 fractions). They will be treated with weekly Gemcitabine (100mg/m2) or daily Nicotinamide (60mg/kg)/Carbogen (2% carbon dioxide, 98% oxygen at 15 litres per minute) if clinically appropriate.

As part of standard treatment patients will have a staging CT scan at diagnosis and a radiotherapy planning CT. Cone beam imaging will also be performed. Response will be assessed as standard with cystoscopy at 3 months and CT scan at 12 months.

As part of the study patients will undergo 4 additional MRI scans. These will take place in the 1st, 2nd, 3rd and 4th weeks of treatment. These MRI scans will include anatomical images - with full and empty bladder as well as cine data (with a scan every minute for 10 minutes) to assess intra fraction motion. They will also include a diffusion weighted imaging (DWI) sequence, which will be used to assess if early prediction of response is possible. The frequency of cone beam imaging will be increased from 6 scans (minimum) as standard of care to 20 scans to allow for daily imaging.

The 1st MRI scan will be contoured to outline the tumour bed, clinical target volumes (CTVs) and OARs. A variety of planning strategies will be developed including standard planning target volume (PTV) margins, a plan of the day (POTD) approach, a POTD+ as well as an online adaptation model. These models will be used to assess coverage of CTV and PTV, and the feasibility of increasing radiation dose to the tumour bed, as well as dose to OARs using the scans obtained during the radiotherapy treatment. The practicality of each approach will also be assessed. Inter and intra fraction organ and tumour bed motion will also be analysed in order to develop patient specific models.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of bladder cancer
* Treatment with primary curative intent
* Undergoing external beam radiotherapy (+/-chemotherapy)
* Age over 18 years

Exclusion Criteria:

* Any contraindications to MRI identified after MRI safety screening including completion of an MRI Safety Screening Form
* Any contraindications to both Hyoscine Butylbromide (Buscopan)
* Previous cystectomy
* Unable to tolerate MRI scans
* Metastatic disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Coverage of the Clinical Target Volume for different adaptive radiotherapy strategies | 18 months
  Coverage of the Clinical Target Volume for different adaptive radiotherapy strategies
Dose to the Organs At Risk for different adaptive radiotherapy strategies | 18 months
  Dose to the Organs At Risk for different adaptive radiotherapy strategies

SECONDARY OUTCOMES:
Diffusion Weighted Imaging on MR prior to and during treatment and clinical response to treatment on post treatment cystoscopy. | 18 months
  Diffusion Weighted Imaging on MR prior to and during treatment and clinical response to treatment on post treatment cystoscopy.
Bladder filling using MR sequences and stratification of patients into large or small bladder and tumour bed motion | 18 months
  Bladder filling using MR sequences and stratification of patients into large or small bladder and tumour bed motion

CONTACTS AND LOCATIONS:
Overall Officials: Ananya Choudhury, MA, PhD, Principal Investigator — The Christie NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No